CLINICAL TRIAL: NCT06380400
Title: The Effect of Foot Bath on Birth Pain and Birth Comfort in the First Stage of Labour
Brief Title: The Effect of Foot Bath on Birth Pain and Birth Comfort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Habibe BAY, Assist prof., Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 0000-0001-5786-4385
Record Dates: First submitted 2024-04-03; First posted 2024-04-23 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Parturition
Keywords: Birth; Labour; Footbath; Birth pain; Birth comfort

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Foot bath intervention group (Experimental): Pregnant women are given a foot bath during the first stage of labour.
  Interventions: Behavioral: Foot bath
- Routine midwifery care control group (No Intervention): Pregnant women receive routine midwifery care during the first stage of labour.

INTERVENTIONS:
Behavioral: Foot bath — Pregnant women were given footbaths for 20 minutes during the active phase of the first stage of labour (after cervical dilatation of 4 cm) and 20 minutes during the transitional phase of the second stage of labour (cervical dilatation of 9 cm). Pregnant women who completed two footbath sessions were assessed for pain using the visual comparison scale. In addition, the data collection process will be completed by applying the Birth Comfort Scale after the two stages of labour.
  Arms: Foot bath intervention group

SUMMARY:
Although childbirth is seen as a natural, happy, meaningful and universal experience, women are often faced with severe pain, discomfort and a sensory state that can be overwhelming. There are two ways to reduce labour pain: pharmacological (drugs) and non-pharmacological (non-drug methods). Non-pharmacological methods, in particular, attempt to relieve pain by addressing emotional, cognitive, behavioural and socio-cultural dimensions. These methods provide relief and reduce the perception of pain. One of the non-pharmacological methods used to reduce labour pain is footbaths. Footbaths are widely used as a nurse/midwife intervention in many countries. Footbathing is a simple technique used to induce a sense of comfort and relaxation. It involves gently immersing the patient's legs and feet (below the knees) in a basin of warm water. Local heat treatments are generally safe and are considered an effective form of complementary medicine. In its simplest form it means "a tool to be part of supportive care, promoting peace, positive emotions, comfort, satisfaction and enjoyment". The mechanisms responsible for the effects of footbathing are not fully understood, but soaking the feet in warm water and stimulating the sense of touch through massage or washing can reduce sympathetic nerve activity, thereby reducing pain and increasing comfort. In other words, reducing pain during labour means providing support and comfort to the woman. This study was designed to evaluate the effect of a foot bath applied in the first stage of labour on labour pain and comfort in nulliparous women.

DETAILED DESCRIPTION:
The purpose of the study will be explained to pregnant women found to meet the inclusion criteria, and written informed consent will be obtained from participants who volunteer for the study. Participants will be randomly divided into two groups (group 1: intervention group, group 2: control group). Pregnant women will be allocated to the intervention and control groups according to the randomisation scheme to be generated from the random.org website. The personal information form will be used for both intervention and control groups.

Intervention group Pregnant women in the intervention group will receive footbaths for 20 minutes during the active phase of the first stage of labour (after 4 cm cervical dilation) and 20 minutes during the transitional phase of the second stage of labour (9 cm cervical dilation). Pregnant women who completed two footbath sessions were assessed for pain using the visual comparison scale. In addition, the data collection process will be completed by applying the birth comfort scale after two stages of labour.

Control group The process of applying the data collection tools to the pregnant women in the control group is the same as for the intervention group. The pregnant women in the control group will be subjected to the routine practices of the hospital without foot bathing.

Warm water foot bath:

The warm water footbath is performed in 4 steps. Before starting the treatment, warm water is poured into the bucket in which the footbath will take place and the water temperature is set at 41-42°C using a thermometer. In the first stage of the application, the room temperature is between 22 and 25°C. In the second stage, the applicants are made to sit in a chair or armchair. In the third stage, they are allowed to dip their feet into the warm water footbath bucket, where the water temperature is kept between 41 and 42°C, up to the level of the ankles. They are asked to remain in this position for 20 minutes. The temperature of the water is checked between applications and hot water is added when the water cools down. At the end of the treatment, the feet are taken out of the water and dried with a towel. The towel should be left on for 5-7 minutes to allow the heat to work for a while.

ELIGIBILITY:
Inclusion Criteria:

* Primipar pregnancy
* 37 and 42 weeks
* Cervical dilation at least 4 cm
* Head presentation
* Over 18 years of age
* Pregnant women who agreed to participate after being informed about the study

Exclusion Criteria:

* People with communication difficulties and mental disabilities
* Any risk condition related to pregnancy (pre-eclampsia, gestational diabetes, anomalies of presentation, anomalies related to the placenta)
* Development of maternal-fetal complications
* Use of anticoagulant therapy
* Pregnant women with a diagnosed psychiatric illness will be excluded from the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Visuell analog scale score of the pregnant woman | within the first 24 hours after the time of the birth of the baby
  Pain levels of pregnant women will be assessed. On one side of the scale there is a line labelled 'no pain' and on the other side there is a line labelled 'severe pain' and on the side immediately behind this line there is a scale divided into 10 equal intervals. The higher the score, the greater the intensity of the pain.

SECONDARY OUTCOMES:
Birth comfort scale score of the pregnant woman | within the first 24 hours after the time of the birth of the baby
  Pregnant women's comfort during childbirth will be assessed. The minimum score that can be obtained from the scale is 14 and the maximum score is 70. The higher the score, the higher the level of comfort.

CONTACTS AND LOCATIONS:
Overall Officials: Habibe Bay Ozcalik, Principal Investigator — Selcuk University
Locations (1):
- Habibe Bay Ozcalik, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Participants' information will not be shared with third parties. Research results will be shared with other researchers after the study is completed